CLINICAL TRIAL: NCT02121184
Title: A Clinical Trial Evaluating the Interaction of Rapid Hydration and the Rate of Oxytocin Labor Augmentation on Fetal Heart Rate Changes and Maternal Fetal Outcomes
Brief Title: Association Between Fluid Administration, Oxytocin Administration, and Fetal Heart Rate Changes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to low enrollment due to competing studies and the PI has now left Northwestern.
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00074673
Record Dates: First submitted 2014-04-16; First posted 2014-04-23 (Estimated); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy; Labor Pain
Keywords: Oxytocin; Labor, Obstetric; Non-reassuring fetal heart rate; Epidural
MeSH Terms: conditions — Labor Pain | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Oxytocin (Active Comparator): Lactated Ringers bolus of 1000 mL will be initiated when the patient is positioned for epidural placement. Oxytocin management will continue as per the routine oxytocin protocol
  Interventions: Drug: Routine oxytocin
- Half-dose Oxytocin (Experimental): Lactated Ringers bolus of 1000 mL will be initiated when the patient is positioned for epidural placement. A half-dose oxytocin will be initiated and not increased until 60 minutes after.
  Interventions: Drug: Half-dose oxytocin

INTERVENTIONS:
Drug: Routine oxytocin — per regular oxytocin protocols
  Other Names: Pitocin
  Arms: Routine Oxytocin
Drug: Half-dose oxytocin — The dose of oxytocin currently being administered will be halved and not increased until after 60 minutes initiation of labor analgesia
  Other Names: Pitocin
  Arms: Half-dose Oxytocin

SUMMARY:
Fetal heart rate patterns are an important parameter in the diagnosis of non-reassuring fetal status. Combined-spinal epidural analgesia is a method of initiating labor analgesia used by approximately 90% of the parturients at Prentice Women's Hospital. Optimizing the variables which could affect fetal heart rate patterns at the time of initiation of analgesia, such as fluid administration and oxytocin management, could help us provide better care for our patients and their fetuses.

Hypotheses: Patients who receive a 1000 mL fluid bolus and lower rates of oxytocin administration will have fewer non-reassuring fetal heart rate (FHR) changes.

DETAILED DESCRIPTION:
Informed, written consent will be obtained. At the time of request for labor analgesia, group assignment will be determined by opening an opaque envelope. Patients will be randomized to one of four groups.

All subjects will receive a maintenance infusion of 125 mL Lactated Ringers (LR) solution throughout the study. For patients in Groups A or B, an intravenous bolus of 1000 mL LR will be initiated when the patient is positioned for epidural placement. The bolus will be administered through a free-flowing wide open intravenous catheter until complete.

Patients in Groups C and D will not receive any additional fluid bolus and will only receive the maintenance infusion of 125 mL LR during the study period. Blinding will be maintained by the Labor and Delivery nurse by covering up the LR bolus fluid bag.

If the patient is randomized to groups B or D, the dose of oxytocin currently being administered will be halved and not increased for the duration of the study period (60 minutes after the initiation of CSE).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Healthy nulliparous or multiparous women
* Term (>36 week gestation)
* Singleton pregnancy
* Spontaneous labor or spontaneous rupture of membranes
* Receive oxytocin
* Request neuraxial analgesia

Exclusion Criteria:

* Under 18 years old
* Presence of any systemic disease (ex: diabetes mellitus, hypertension, preeclampsia
* Use of chronic analgesic medications
* Prior administration of system opioid labor analgesia
* Non-vertex presentation
* Induction of Labor
* Contraindication to neuraxial analgesia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hogue, M.D., Study Chair — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mardirosoff C, Dumont L, Boulvain M, Tramer MR. Fetal bradycardia due to intrathecal opioids for labour analgesia: a systematic review. BJOG. 2002 Mar;109(3):274-81. doi: 10.1111/j.1471-0528.2002.01380.x. PMID 11950182
- [Background] Abrao KC, Francisco RPV, Miyadahira S, Cicarelli DD, Zugaib M. Elevation of uterine basal tone and fetal heart rate abnormalities after labor analgesia: a randomized controlled trial. Obstet Gynecol. 2009 Jan;113(1):41-47. doi: 10.1097/AOG.0b013e31818f5eb6. PMID 19104358
- [Background] Clarke VT, Smiley RM, Finster M. Uterine hyperactivity after intrathecal injection of fentanyl for analgesia during labor: a cause of fetal bradycardia? Anesthesiology. 1994 Oct;81(4):1083. doi: 10.1097/00000542-199410000-00041. No abstract available. PMID 7943823
- [Background] Lopez-Zeno JA, Peaceman AM, Adashek JA, Socol ML. A controlled trial of a program for the active management of labor. N Engl J Med. 1992 Feb 13;326(7):450-4. doi: 10.1056/NEJM199202133260705. PMID 1732771
- [Background] Lindmark G, Nilsson BA. A comparative study of uterine activity in labour induced with prostaglandin F2alpha or oxytocin and in spontaneous labour. I. Pattern of the uterine contractions. Acta Obstet Gynecol Scand. 1976;55(5):453-60. doi: 10.3109/00016347609158529. PMID 998176
- [Background] Satin AJ, Leveno KJ, Sherman ML, Brewster DS, Cunningham FG. High- versus low-dose oxytocin for labor stimulation. Obstet Gynecol. 1992 Jul;80(1):111-6. PMID 1603479
- [Background] Hourvitz A, Alcalay M, Korach J, Lusky A, Barkai G, Seidman DS. A prospective study of high- versus low-dose oxytocin for induction of labor. Acta Obstet Gynecol Scand. 1996 Aug;75(7):636-41. doi: 10.3109/00016349609054688. PMID 8822656
- [Background] Merrill DC, Zlatnik FJ. Randomized, double-masked comparison of oxytocin dosage in induction and augmentation of labor. Obstet Gynecol. 1999 Sep;94(3):455-63. doi: 10.1016/s0029-7844(99)00338-5. PMID 10472877
- [Background] Sadler LC, Davison T, McCowan LM. A randomised controlled trial and meta-analysis of active management of labour. BJOG. 2000 Jul;107(7):909-15. doi: 10.1111/j.1471-0528.2000.tb11091.x. PMID 10901564
- [Background] Kinsella SM, Pirlet M, Mills MS, Tuckey JP, Thomas TA. Randomized study of intravenous fluid preload before epidural analgesia during labour. Br J Anaesth. 2000 Aug;85(2):311-3. doi: 10.1093/bja/85.2.311. PMID 10992845
- [Background] Cheek TG, Samuels P, Miller F, Tobin M, Gutsche BB. Normal saline i.v. fluid load decreases uterine activity in active labour. Br J Anaesth. 1996 Nov;77(5):632-5. doi: 10.1093/bja/77.5.632. PMID 8957980
- [Background] ACOG Practice Bulletin No. 106: Intrapartum fetal heart rate monitoring: nomenclature, interpretation, and general management principles. Obstet Gynecol. 2009 Jul;114(1):192-202. doi: 10.1097/AOG.0b013e3181aef106. No abstract available. PMID 19546798

RESULTS

PARTICIPANT FLOW:
Groups:
- Half- Dose Oxytocin: Lactated Ringers bolus of 1000 mL will be initiated when the patient is positioned for epidural placement. A half-dose oxytocin will be initiated and not increased until 60 minutes after.
  Half-dose oxytocin: The dose of oxytocin currently being administered will be halved and not increased until after 60 minutes initiation of labor analgesia
Period: Overall Study
Arm/Group | Routine Oxytocin | Half- Dose Oxytocin
Started | 86 | 86
Completed | 84 | 83
Not Completed | 2 | 3
Not completed — No oxytoxin administered prior to combined spinal epidural catheter placement | 1 | 0
Not completed — Multiple parasthesias at time after combined spinal epidural catheter placement | 0 | 1
Not completed — Emergency cesarean section required | 0 | 2
Not completed — Combined spinal epidural completed without notifying study team | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Lactated Ringers bolus of 1000 mL will be initiated when the patient is positioned for epidural placement. Oxytocin management will continue as per the routine oxytocin protocol
  Routine oxytocin: per regular oxytocin protocols
- Group B: Lactated Ringers bolus of 1000 mL will be initiated when the patient is positioned for epidural placement. A half-dose oxytocin will be initiated and not increased until 60 minutes after.
  Half-dose oxytocin: The dose of oxytocin currently being administered will be halved and not increased until after 60 minutes initiation of labor analgesia
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Continuous [Mean (Full Range); unit: Years] | 32.9 [19 to 44] | 32.35 [23 to 43] | 32.5 [19 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 86 | 172
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 83 | 77 | 160
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 14 | 24
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 5 | 16
  White | 58 | 56 | 114
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 11 | 17
Fetus gestational age in weeks [Mean (Full Range); unit: Weeks] | 39 [37.4 to 40.3] | 39.3 [37.5 to 40.5] | 39.1 [37.4 to 40.5]
Maternal weight [Mean (Full Range); unit: Kilograms] | 80.31 [60.2 to 170] | 79.26 [57.1 to 136.8] | 79.7 [57.1 to 170]
Maternal Mean Arterial Pressure [Mean (Full Range); unit: millimeters mercury] — Mean arterial pressure equals diastolic pressure + 1/3 (systolic pressure - diastolic pressure)
  millimeters mercury | 92.06 [52 to 111] | 89.94 [72 to 111] | 91.07 [52 to 111]
Oxytocin dose at start of epidural procedure [Mean (Full Range); unit: milliunits/mL] — Oxytocin dose milliunits/mL is administered via intravenous catheter.
  milliunits/mL | 7.39 [0 to 22] | 8.38 [0 to 18] | 7.9 [0 to 22]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Non-reassuring Fetal Heart Rate Tracings.
Description: Incidence of non-reassuring fetal heart rate tracings during the first 60 minutes after the placement of epidural analgesia
Time Frame: Request for labor analgesia up to the first 60 minutes after the epidural placement
Population: Data was not collected as the OB/MD who was a certified fetal heart rate evaluator on the team (OB/MD) left Northwestern University. The fetal heart rate data can only be collected, scored and analyzed by a certified fetal heart rate evaluator and there are none available for this project.
Arm/Group | Routine Oxytocin | Half-dose Oxytocin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 7 days after study intervention.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 0/86 | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=86) | Group B (N=86)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) — Nausea

LIMITATIONS AND CAVEATS:
Ended trial early due to low enrollment. Could not obtain a certified assessments of fetal heart tracings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT02121184/Prot_SAP_000.pdf